CLINICAL TRIAL: NCT03024645
Title: Be a Mom: A Randomized Controlled Trial of the Effectiveness of a Web-based Preventive Intervention for Postpartum Depression.
Brief Title: Be a Mom: Effectiveness of a Web-based Preventive Intervention for Postpartum Depression
Acronym: BeAMom
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Ana Fonseca, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CINEICC-2-BaM; SFRH/BPD/93996/2013 (Other Grant/Funding Number: Portuguese Scientific Foundation)
Record Dates: First submitted 2016-12-19; First posted 2017-01-19 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: PostPartum Depression
Keywords: Postpartum Depression; Cognitive-Behavioral Therapy; Prevention; Web-Based Psychological Intervention
MeSH Terms: conditions — Depression, Postpartum | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BeAMom (Experimental): High-risk (HR) women will receive a web-based preventive intervention for PPD (the Be a Mom program). In addition, women will receive postpartum and and pediatric treatment as usually performed in primary care settings (TAU).
  Interventions: Behavioral: Be A Mom; Other: Treatment as usually (TAU)
- Control (Active Comparator): High-risk (HR) women will receive postpartum and pediatric treatment as usually performed in primary care settings (TAU). During medical appointments, health professionals may ask women and provide information about psychological problems during the postpartum period.
  Interventions: Other: Treatment as usually (TAU)

INTERVENTIONS:
Behavioral: Be A Mom — The Be a Mom program is a web-based self-guided cognitive-behavioral intervention to prevent postpartum depression, targeting postpartum women. It consists of 5 weekly modules, each module targeting a specific thematic content, and providing women with both information and specific therapeutic strategies (with a strong focus on cognitive-behavioral techniques) to address each thematic content. Modules are sequential.
  Arms: BeAMom
Other: Treatment as usually (TAU) — performed in primary care settings

SUMMARY:
The main goal of the research is to apply and evaluate the web-based preventive intervention (the Be a Mom program), in terms of its efficacy, acceptability and feasibility (user's adherence, dropout), and user's satisfaction. Prior to the randomized controlled trial (RCT), the investigators will conduct a pilot trial to evaluate the preliminary version of the Be a Mom program in high-risk women (random assignment to the intervention or to the control condition).

The RCT will be a two-arm prevention trial. Women who have had a child during the prior month will be enrolled in the study. A minimum number of 1000 women will be enrolled in the study. After agreeing to participate in the study, the women will be screened for the presence of risk factors for PPD and early-onset PPD symptoms (using self-report questionnaires) by a researcher (licensed psychologist). In case of a negative screen, women's participation in the study will end. In case of a positive screen (high-risk women), women will be randomly assigned to one of the conditions: the intervention (Be a Mom program) or the control condition. The sample will be recruited online and at the maternities of Coimbra University Hospitals-CHUC, EPE.

Participation in the study will last 11 months. The Be a Mom program will last 5 weeks. Participants in both conditions will be invited by the researchers via email to complete baseline, post-intervention and follow-up (4-months and 12-months after childbirth) assessments. Assessments will include self-report questionnaires to assess several indicators (e.g., depressive and anxiety symptoms, dyadic adjustment, mother-child bonding, and maternal confidence), mechanisms that may be involved in the treatment response (e.g., npsychological flexibility, emotional regulation) and user's acceptability and satisfaction.

DETAILED DESCRIPTION:
In the present study, a web-based intervention to prevent PPD (the Be a Mom program) will be tested. The design and content development of the Be a Mom program was conducted through a formative evaluation process (including a systematic literature review about the characteristic and content of existing effective preventive interventions for PPD and a focus group with stakeholders to identify the perceived needs of the target population.

Be a Mom is self-guided intervention grounded on CBT principles, and besides addressing the key topics in the prevention of depression, it also addresses key content areas that are associated with risk for PPD (e.g., communication skills that may help women to manage the transition to motherhood). Moreover, it also includes recent developments in acceptance and commitment based-therapies, specifically for the perinatal context. Be a Mom has a modular set-up that is updated weekly, with each module addressing one or two specific thematic contents (Changes and reorganizations during the transition to parenthood; Emotional diversity; Cognitions; Relationship with others [social support and communication]; Couple relationship; Signs and symptoms of depression and help-seeking). In each module, participants will be provided with both psychoeducational content and therapeutic strategies. Informational material will be given in text format, combined with audio, video and/or animations. The Be a Mom program will also include interactive tools and feedback tools to support learning.

The Be a Mom program will be delivered during the postpartum period, as this was identified as privileged time for the implementation of preventive approaches for PPD. Moreover, the Be a Mom program is recommended to target high-risk women (i.e., women who present antenatally identified risk factors for PPD or with early-onset depressive symptoms).

The main goal of the research is to apply and evaluate the web-based preventive intervention (the Be a Mom program), in terms of its efficacy, acceptability and feasibility (user's adherence, dropout), and user's satisfaction. The efficacy of the program will be assessed considering two indicators: a) absence of clinically significant depressive symptoms at post-intervention and throughout the first postpartum year; and b) post-intervention and follow-up improvements in mother's psychosocial adjustment indicators (anxiety symptoms, maternal confidence and dyadic adjustment). The present study will also aim to investigate the mechanisms explaining the treatment response (e.g., negative automatic thoughts, psychological flexibility, self-compassion).

The research design of the trial followed the methodological recommendations for the development and evaluation of web-based interventions. Prior to the randomized controlled trial (RCT), a pilot trial to evaluate the preliminary version of the Be a Mom program will be conducted. The pilot study will be conducted with women presenting high-risk for PPD or early-onset depressive symptoms (assessed one-month postpartum through self-report questionnaires). The investigators will randomly assign high-risk women to the intervention (the Be a Mom program) or to the control condition, and women will be assessed at baseline and post-intervention concerning adjustment outcomes, acceptability, feasibility and user's satisfaction. After completing the assessments, the control group will be provided with the Be a Mom program. The sample will be collected at the Maternity Daniel de Matos and Maternity Bissaya Barreto (both maternities of Coimbra University Hospitals -CHUC, EPE) and online. Data collection methods will include several self-administered questionnaires. Based on research results the modifications will be identified and conducted to develop the final version of the Be a Mom program, allowing for further efficacy studies.

The RCT will be a two-arm prevention trial, conducted in high-risk women (i.e., presenting risk factors for PPD and/or early-onset postpartum depressive symptoms). The intervention condition (the Be a Mom program) will be compared with a control condition (Treatment as Usual). The sample will include women who delivered an healthy baby in the early postpartum period (up to 3 months postpartum). Women will be enrolled both online and at the maternities of Coimbra University Hospitals -CHUC, EPE. A minimum number of 150 women per condition will be required (N=300). Accounting for the proportion of high-risk and low-risk women and the 50% of attrition rate over time, an anticipated sample of 1000 women will be enrolled in the study.

A researcher (licensed psychologist) will conduct an interview with women who demonstrate interest in the study, aiming to explain the study goals, the structure and arms of the research and the researchers' and participants' roles. Women who agree to participate in the study will sign an informed consent form. All ethical requirements for research with humans are guaranteed.

After women's agreement to participate in the study, the researcher (licensed psychologist) will screen women for the presence of risk factors for PPD and early-onset PPD symptoms (using self-report questionnaires). In case of a negative screen, women's participation in the study will end. In case of a positive screen, high-risk women will be randomly assigned (blocked randomization, with allocation concealment) to one of the conditions: the intervention (Be a Mom program) or the control condition. The randomization will be conducted by a different researcher who will be blind to the assessment procedure.

Participation in the study will last 11 months. The Be a Mom program will last 5 weeks. Participants in both conditions will be invited via email to complete baseline, post-intervention and follow-up (4-months and 12-months after childbirth) assessments. Assessments will include self-report questionnaires to assess several indicators (e.g., depressive and anxiety symptoms, dyadic adjustment, mother-child bonding, and maternal confidence), mechanisms that may be involved in the treatment response (e.g., psychological flexibility, emotional regulation) and user's acceptability and satisfaction. The necessary statistical analyses will be conducted, using the intention-to-treat principles.

ELIGIBILITY:
General Inclusion Criteria:

* Having 18 years or more (being an adult);
* Being female;
* Having had a live healthy birth in the last women, with both women and the child discharged from hospital;
* Home access to the internet.

Inclusion criteria for the High-Risk women group (to continue the participation in the study):

* Presence of risk factors for PPD (PDPI-R ≥ 5.5) and/or early-onset depressive symptoms (EPDS > 9);

Exclusion Criteria:

* Current diagnosis of serious mental health condition (substance abuse, bipolar disorder);
* Currently receiving treatment for depressive symptoms, including antidepressant medication or psychotherapy;
* Language difficulties that impede comprehension/reading-writing;

All participants will be informed that they will be randomized to one of the study groups and that will only be included if they give informed consent to participate in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of women with clinically significant postpartum depressive symptoms (EPDS > 12) at 4 months postpartum | 4 months postpartum
  Measured with EPDS
Number of women with clinically significant postpartum depressive symptoms (EPDS > 12) at 12 months postpartum | 12 months postpartum
  Measured with EPDS
Changes from baseline in the severity of depressive symptoms | From baseline to 12 months postpartum
  Measured with EPDS

SECONDARY OUTCOMES:
Changes from baseline in anxiety symptoms | From baseline to 12 months postpartum
  Measured with Anxiety Subscale of HADS
Changes from baseline in quality of life | From baseline to 12 months postpartum
  Measured with EQ-5D
Changes from baseline in dyadic adjustment | From baseline to 12 months postpartum
  Measured with Dyadic Adjustment Scale - Revised
Changes from baseline in maternal confidence | From baseline to 12 months postpartum
  Measured with the Parental Confidence Questionnaire
Changes from baseline in the frequency of negative automatic thoughts | From baseline to 12 months postpartum
  Measured with the Postnatal Negative Thoughts Questionnaire
Changes from baseline in psychological flexibility | From baseline to 12 months postpartum
  Measured with the Acceptance and Action Questionnaire-II
Changes from baseline in self-criticism and self-compassion | From baseline to 12 months postpartum
  Measured with the Self-Compassion Scale (short form)
Changes from baseline in emotional regulation | From baseline to 12 months postpartum
  Measured with the Difficulties in Emotional Regulation Scale
Acceptability of the program for postpartum women | Measured at post-intervention (2,5 months postpartum)
  Measured through specific questions (to be developed by the researchers) to assess acceptability.
Feasibility of the program for postpartum women as measured by number of website logins | Measured at post-intervention (2,5 months postpartum).
  Measured through the number of user's website logins.
Feasibility of the program for postpartum women as measured by website average visit length | Measured at post-intervention (2,5 months postpartum).
  Measured through the number of user's website average visit length.
Feasibility of the program for postpartum women as measured by number of exercises completed | Measured at post-intervention (2,5 months postpartum).
  Measured through the total number of exercises completed by the users.
Feasibility of the program for postpartum women as measured by dropout rate. | Measured at post-intervention (2,5 months postpartum).
  Measured through the number of users that dropped out from the web-based intervention before completing it.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Fonseca, PhD, Principal Investigator — Post-doctoral fellow at CINEICC
Locations (1):
- Ana Fonseca, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
After the conclusion of the trial, the investigators plan to share the results of the study both with scientific community and health professionals.

REFERENCES:
- [Background] Fonseca, A., Pereira, M., Araújo-Pedrosa, A., Gorayeb, R., & Canavarro, M. C. (2016, november). Web-based preventive intervention for postpartum depression: Development and formative evaluation of a CBT intervention. Poster presented at the IX International Congress and XIV National Congress in Clinical Psychology, Santander, Spain. https://www.researchgate.net/publication/311733757_Web-based_preventive_intervention_for_postpartum_depression_Development_and_formative_evaluation_of_a_CBT_intervention
- [Background] Fonseca, A., Pereira, M., Araújo-Pedrosa, A., Moura-Ramos, M., Gorayeb, R., & Canavarro, M. C. (in press). Be a Mom: Formative evaluation of a web-based psychological intervention to prevent postpartum depression. Cognitive and Behavioral Practice. doi:10.1016/j.cbpra.2018.02.002
- [Derived] Carona C, Pereira M, Araujo-Pedrosa A, Canavarro MC, Fonseca A. The Efficacy of Be a Mom, a Web-Based Intervention to Prevent Postpartum Depression: Examining Mechanisms of Change in a Randomized Controlled Trial. JMIR Ment Health. 2023 Mar 17;10:e39253. doi: 10.2196/39253. PMID 36930182